CLINICAL TRIAL: NCT03491423
Title: Short and Fast Step Test: Feasibility, Validity and Tolerance of a Functional Evaluation Test of Lactic Anaerobic Capacities in Patients With Coronary Artery Disease
Acronym: CORANAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HANNEQUIN APPARA 2016
Record Dates: First submitted 2018-03-30; First posted 2018-04-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease Without Heart Failure
MeSH Terms: interventions — epicatechin gallate; Heart Rate; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: Short and fast step test without measurement of pulmonary gas exchange; Biological: glucose meter; Other: ECG / heart rate; Other: questionnaires; Other: Short and fast step test with measurement of pulmonary gas exchange

INTERVENTIONS:
Other: Short and fast step test without measurement of pulmonary gas exchange — For one minute, the patient should climb up and down a 17.5 cm high step as quickly as possible while holding onto a bar in front of the step.
Biological: glucose meter — glucose meter to measure lactatemia
Other: ECG / heart rate — ECG and heart rate (HR) collection by telemetry
Other: questionnaires — VAS pain assessment and evaluation of effort perception according to Borg's scale
Other: Short and fast step test with measurement of pulmonary gas exchange — For one minute, the patient should climb up and down a 17.5 cm high step as quickly as possible while holding onto a bar in front of the step.

SUMMARY:
Recommendations for cardiovascular rehabilitation (CVR) encourage exercise training, primarily involving the aerobic system, to allow patients to regain independence in daily activities. However, the lactic anaerobic process is also involved during these activities (stair climbing, carrying loads, etc.). Hence there is a major interest in accurately assessing patients' anaerobic capacities in order to tailor suitable exercise programs. However, there are no functional tests specifically dedicated to the evaluation of lactic anaerobic metabolism and adapted to people with coronary disease. The investigators offer a dedicated test, the short and fast test (SFST), which can be applied in current clinical practice and has already been evaluated in a population of healthy subjects. The purpose of this project is to evaluate the safety, feasibility and validity of SFST in a population of patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

- Patient who has given oral consent Adult patient (male or female) with coronary artery disease without heart failure referred for rehabilitation program Left ventricular ejection fraction (Simpson method) > 45%.

Exclusion Criteria:

* Protected adult
* Patient not affiliated to a national health insurance scheme
* Pregnant or breastfeeding woman
* Orthostatic hypotension
* Severe obstructive heart disease
* aortic valve narrowing
* Progressive severe cardiac rhythm or conduction disorders not requiring a device, detected during the initial stress test.
* intracavitary cardiac thrombus
* severe pulmonary arterial hypertension (systolic pulmonary hypertension >70mmHg)
* recent venous thromboembolic history (last 3 months)
* heart transplantation
* associated medical condition that can predominantly impair functional and respiratory capacities (examples: unstabilized metabolic disorders such as progressive renal failure, significant asthenia related to a severe unstabilized condition such as neoplasia, systemic disease, chronic obstructive pulmonary disease...)
* physical impairments of the lower limbs hindering the test, whether neurological (central or peripheral), arterial (in particular, arteriopathy of the lower limbs with systolic index < 0.6) or orthopedic (degenerative or inflammatory rheumatism)
* Treatment with Corticosteroids, Anabolics, or L-Carnitine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
percentage of patients who completed the SFST without complications | through study completion, an average of 11 days
  - Absence of muscular or bone-joint disorders quantified according to the VAS. The exercise will be considered as not tolerated if pain is reported during the test and/or at day 3 (VAS≥6).
  AND no falls or stumbling related trauma
  AND absence of cardiovascular or blood pressure events:
  * Hypertension (systolic pressure greater than 250 mmHg (O'Brien et al. 2005) or hypotension with clinical consequences (malaise or feeling unwell)
  * Discomfort, chest pain, onset of vascular claudication
  * Rhythm or conduction disorders or repolarization abnormalities, at a higher frequency than that observed in the pre-inclusion stress test
  * Abnormal increase in heart rate (greater than the maximum rate determined during the stress test).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Result] Besson D, Gouteron A, Sinssaine-Ayillo A, Casillas JM, Rigaud L, Ornetti P, Fournel I, Ksiazek E, Laroche D, Gueugnon M. Is the Short and Fast Step Test a safe and feasible tool for exploring anaerobic capacities of individuals with coronary heart disease in clinical practice? Eur J Phys Rehabil Med. 2021 Dec;57(6):977-984. doi: 10.23736/S1973-9087.21.06713-7. Epub 2021 Feb 23. PMID 33619946